CLINICAL TRIAL: NCT05730933
Title: An Intervention Study to Improve Therapeutic Compliance in Adult Patients With Eosinophilic Esophagitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. A.J. (Arjan) Bredenoord, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL82384.018.22
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis; maintenance treatment; compliance; intervention
MeSH Terms: conditions — Eosinophilic Esophagitis; Patient Compliance | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Intervention — Subjects will receive a behavioral intervention with additional education in combination with more frequent follow up and patient reminders
  Arms: Intervention

SUMMARY:
In many chronic conditions adherence to long-term treatment is a challenge, also for patients with eosinophilic esophagitis. Interventions, such as behavioral, educational and reminder interventions might improve treatment adherence. With this trial the investigators want to assess the effects of additional education in combination with more frequent follow up and patient reminders on adherence to treatment in adult patients with eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female patient
* Age >18 years
* Previous diagnosis of EoE, confirmed by histopathology, with the presence of >15 eosinophilic granulocytes per high power field (hpf) in esophageal biopsies
* Current maintenance treatment for EoE with a PPI or swallowed topical corticosteroids or about to start with these maintenance medications as decided during regular clinical practice

Exclusion Criteria:

* Severe and clinically unstable concomitant disease that may interfere with the subject's ability to participate in the study
* Receive investigational treatment during the study
* Dilation of esophagus required
* Insufficient Dutch or English language skills to understand patient information leaflets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence at 12 weeks | 12 weeks
  Treatment adherence, defined as the proportion of subjects in both groups that meet a desired adherence rate of > 80%, calculated by pill count adherence rate

SECONDARY OUTCOMES:
Treatment adherence at 6 months | 6 months
  Treatment adherence, defined as the proportion of subjects in both groups that meet a desired adherence rate of > 80%, calculated by pill count adherence rate
Treatment adherence at 12 months | 12 months
  Treatment adherence, defined as the proportion of subjects in both groups that meet a desired adherence rate of > 80%, calculated by pill count adherence rate
Differences in self-reported treatment adherence measured by brief-IPQ | 12 weeks, 6 months and 12 months.
  Differences in self-reported treatment adherence measured by brief-IPQ, a 9 item questionnaire where every item is assessed individually (0 to 10 response scale) except for 1 open-ended response item
Differences in self-reported treatment adherence measured by BMQ | 12 weeks, 6 months and 12 months.
  Differences in self-reported treatment adherence measured by BMQ, questionnaire with 2 subscales. Necessity subscale ranges from 5-20, where lower scores indicate low necessity beliefs. Concern scale ranges from 5-20 where lower scores indicate higher confidence in positive effects of medication.
Differences in self-reported treatment adherence measured by 8-point MMAS | 12 weeks, 6 months and 12 months.
  Differences in self-reported treatment adherence measured by 8-point MMAS. Total scores range between 0 to 8, where a higher score indicates higher treatment adherence
Differences in self-reported treatment adherence measured by MARS questionnaire | 12 weeks, 6 months and 12 months.
  Differences in self-reported treatment adherence measured by MARS questionnaire 5. Scores range between 1-25, where a higher score indicates higher reported treatment adherence
Change in clinical symptoms measured by DSQ questionnaire | 12 weeks, 6 months and 12 months
  Change in clinical symptoms measured by DSQ questionnaire. Total score range from 0 to 84, where higher scores indicate more symptoms
Change in clinical symptoms measured by SDI questionnaire | 12 weeks, 6 months and 12 months
  Change in clinical symptoms measured by SDI questionnaire. Total scores of the SDI ranges between 0 to 9, where higher scores indicate more symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No